CLINICAL TRIAL: NCT01040143
Title: A Study to Assess the Impact of Pneumococcal Conjugate Vaccination Programme on the Carriage of Pneumococci
Acronym: Pneucast
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Professor Elizabeth Miller, Health Protection Agency
Other Study IDs: PneuCaSt
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2010-09

CONDITIONS: Pneumococcal Disease
Keywords: Pneumococci; Streptococcus pneumoniae
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
A study taking swabs from the back of the nose (nasopharynx) to look at carriage of pneumococci.

ELIGIBILITY:
Inclusion Criteria:

* Born in a cohort eligible for routine or catch up pneumococcal conjugate vaccination (i.e. date of birth since 4th September 2004) or a family member where a child is eligible and has been enrolled
* Written informed consent given by the subject's parent/ legal guardian as well as assent from the child after the nature of the study has been explained to them or
* Written informed consent given by the subject after the nature of the study has been explained to them

Exclusion Criteria:

* Moderate to severe disability.
* Cerebral palsy, syndromes and neurological disorders affecting swallowing.
* Ear Nose and Throat disorders affecting the anatomy of the ear,i.e.malformed ears.
* Confirmed or suspected immunodeficiency (congenital or acquired).
* On immunosuppressive therapy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community samples taken within the home of eligible subjects.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Presence of pneumococci in nasopharyngeal swabs

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Health Protection Agency, Stevenage, Hertfordshire
  - Health Protection Agency, Gloucester
  - Health Protection Agency, London

REFERENCES:
- [Result] van Hoek AJ, Sheppard CL, Andrews NJ, Waight PA, Slack MP, Harrison TG, Ladhani SN, Miller E. Pneumococcal carriage in children and adults two years after introduction of the thirteen valent pneumococcal conjugate vaccine in England. Vaccine. 2014 Jul 23;32(34):4349-55. doi: 10.1016/j.vaccine.2014.03.017. Epub 2014 Mar 21. PMID 24657717
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/24657717